CLINICAL TRIAL: NCT04771845
Title: Transcranial Magnetic Stimulation (TMS) in Patients With Mild Cognitive Impairment (MCI) and Alzheimer Disease (AD): A Twelve-year Retrospective Observational Study
Brief Title: Transcranial Magnetic Stimulation in Mild Cognitive Impairment and Alzheimer Disease
Status: Completed | Type: Observational
Sponsor: The New York Memory Services (Other)
Responsible Party: Principal Investigator, Gayatri Devi, MD, Principal Investigator, The New York Memory Services
Other Study IDs: 20-0812
Record Dates: First submitted 2021-02-07; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: TMS; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- EEG-grid-guided-TMS: Patients with Alzheimer disease and mild cognitive impairment receiving TMS using electroencephalogram grid guided navigation
  Interventions: Device: Transcranial Magnetic Stimulation
- MRI-guided-TMS: Patients with Alzheimer disease and mild cognitive impairment receiving TMS using MRI guided navigation
  Interventions: Device: Transcranial Magnetic Stimulation
- NACC controls: National Alzheimer's Coordinating Center matched controls

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Magnetic stimulation to alter neural activity
  Other Names: TMS
  Groups: EEG-grid-guided-TMS; MRI-guided-TMS

SUMMARY:
The investigators reviewed 12 years of clinical use in an outpatient neurology setting of transcranial magnetic stimulation (TMS) in patients with Alzheimer's disease (AD) and mild cognitive impairment (MCI) to evaluate safety and efficacy of TMS.

DETAILED DESCRIPTION:
The investigators compiled demographic, clinical, and neurocognitive data on all patients who had received TMS for any reason in the clinic over a 12-year period. Of 236 patients receiving TMS, 59 patients with AD and 14 with MCI satisfied study criteria and were compared to controls from the National Alzheimer's Coordinating Center (NACC). Neurocognitive outcomes were compared between magnetic resonance imaging (MRI) and electroencephalogram (EEG)-grid guided TMS in patients. Tolerability data was reviewed for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the National Institute of Neurological and Communicative Disorders and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS- ADRDA) criteria for possible or probable Alzheimer's disease.
* Patients meeting the National Institute of Neurological and Communicative Disorders and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS- ADRDA) criteria for mild cognitive impairment.
* Patients must have undergone at least two standardized neurocognitive batteries before and after beginning TMS.
* Patients must have received greater than or equal to five (5) TMS sessions in less than one year.

Exclusion Criteria:

• Patients with dementias from other causes, such as Lewy Body disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer disease or mild cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Controlled Oral Word Association Test | 05/01/2008-05/30/2020
  Animal score and percentile
Boston 30-item naming test | 05/01/2008-05/30/2020
  spontaneous correct (without cues)
Boston 30-item naming test | 05/01/2008-05/30/2020
  total correct (with cues)
Wechsler Adult Intelligence Scale III | 05/01/2008-05/30/2020
  Digit span
Wechsler Adult Intelligence Scale III | 05/01/2008-05/30/2020
  verbal quotient score and percentile
Wechsler Adult Intelligence Scale III | 05/01/2008-05/30/2020
  performance quotient score and percentile
Wechsler Adult Intelligence Scale III | 05/01/2008-05/30/2020
  object assembly
Wechsler Memory Scale III | 05/01/2008-05/30/2020
  Immediate memory score and percentile
Wechsler Memory Scale III | 05/01/2008-05/30/2020
  Auditory delayed memory score and percentile
Wechsler Memory Scale III | 05/01/2008-05/30/2020
  Visual delayed memory score and percentile
Buschke Selective Reminding Test, 12 item | 05/01/2008-05/30/2020
  Total recall score
Buschke Selective Reminding Test, 12 item, 15 minute | 05/01/2008-05/30/2020
  Delayed recall score
Rosen Drawing Test | 05/01/2008-05/30/2020
  Total score
Processing speed | 05/01/2008-05/30/2020
  Total score and percentile
Mini-mental status examination | 05/01/2008-05/30/2020
  Total score

CONTACTS AND LOCATIONS:
Overall Officials: Gayatri Devi, MD, Principal Investigator — NY Memory

IPD SHARING:
Plan to Share IPD: No